CLINICAL TRIAL: NCT00074165
Title: A Phase II Trial Involving Patients With Recurrent PCNSL Treated With Carboplatin/BBBD, by Adding Rituxan (Rituximab), An Anti CD-20 Antibody, To The Treatment Regimen
Brief Title: Treating Patients With Recurrent PCNSL With Carboplatin/BBBD and Adding Rituxan To The Treatment Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000641; 5R01CA137488-15 (NIH); ONC-02059-LX (Other: OHSU Knight Cancer Institute); 641 (Other: OHSU eIRB); 7465 (Other: OHSU IRB (discontinued number)); OHSU-641 (Other: OHSU IRB); NCT00261651 (obsolete NCT alias)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2011-11-16 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Brain and Central Nervous System Tumors; Drug/Agent Toxicity by Tissue/Organ; Lymphoma; Thrombocytopenia
Keywords: drug/agent toxicity by tissue/organ; thrombocytopenia; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Drug-Related Side Effects and Adverse Reactions; Lymphoma; Thrombocytopenia; Intraocular Lymphoma | interventions — Rituximab; Cyclophosphamide; Etoposide; etoposide phosphate; Carboplatin; sodium thiosulfate; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental)
  Interventions: Drug: Rituxan; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Etoposide phosphate; Drug: Carboplatin; Drug: Sodium thiosulfate; Drug: Neupogen; Drug: Neulasta; Drug: Cytarabine

INTERVENTIONS:
Drug: Rituxan — Total dose: 375mg/m2 infused IV; Every 4 weeks for up to one year.
  Other Names: Rituximab
Drug: Cyclophosphamide — Dose 330mg/m2 x 2 days infused IV; Every 4 weeks for up to 1 year
Drug: Etoposide — Dose 200mg/m2 x 2 days infused IV; Every 4 weeks for up to one year. Etoposide phosphate may be given instead.
Drug: Etoposide phosphate — Dose 200mg/m2 infused IV x 2 days; Every 4 weeks for up to one year. Etoposide may be given instead.
Drug: Carboplatin — Dose: 200mg/m2 x 2 days infused IA with BBBD; Every 4 weeks for up to one year.
Drug: Sodium thiosulfate — Dose: 4 hrs post carboplatin = 20gm/m2;
  Dose: 8 hrs post carboplatin = 16gm/m2
  Infused IV x 2 days
  Other Names: STS
Drug: Neupogen — 48 hours after chemotherapy, QD x 7-10 days until WBC greater than 5000. Neulasta (Pegfilgrastim) may be given instead.
  Other Names: G-CSF; filgrastim
Drug: Neulasta — Dose: 6mg, 24-72 hours after chemotherapy. Neupogen may be given instead.
  Other Names: Pegfilgrastim
Drug: Cytarabine — Dose: 40mg on Day 14 following chemotherapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as carboplatin, cyclophosphamide, etoposide, etoposide phosphate, and cytarabine, use different ways to stop cancer cells from dividing so they stop growing or die. Osmotic blood-brain barrier disruption uses certain drugs to open the blood vessels around the brain and allow anticancer substances to be delivered directly to the brain tumor. Chemoprotective drugs such as sodium thiosulfate may protect normal cells from the side effects of carboplatin-based chemotherapy. Combining rituximab with chemotherapy given with osmotic blood-brain barrier disruption plus sodium thiosulfate may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining rituximab with combination chemotherapy given with osmotic blood-brain barrier disruption plus sodium thiosulfate in treating patients who have refractory or recurrent primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of rituximab, carboplatin, cyclophosphamide, etoposide or etoposide phosphate and cytarabine administered in conjunction with osmotic blood-brain barrier disruption and high-dose sodium thiosulfate, in terms of complete response rate, in patients with refractory or recurrent primary CNS lymphoma.

Secondary

* Determine the overall survival and 2-year progression-free survival of patients treated with this regimen.
* Determine the quality of life and cognitive function of patients treated with this regimen.
* Determine the neurotoxicity of this regimen in these patients.
* Determine the percentage of patients with ototoxicity over time after treatment with this regimen.
* Determine the effect of delayed administration of sodium thiosulfate on granulocyte and erythrocyte counts in these patients.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on day 1. On days 2 and 3, patients receive carboplatin intra-arterially over 10 minutes, cyclophosphamide IV over 10 minutes, and etoposide or etoposide phosphate IV over 10 minutes in conjunction with blood-brain barrier disruption. Patients also receive high-dose sodium thiosulfate IV over 15 minutes administered 4 and 8 hours after carboplatin on days 2 and 3 and intraventricular or intrathecal cytarabine on day 14. Beginning 48 hours after the last dose of chemotherapy, patients receive filgrastim (G-CSF)* subcutaneously (SC) daily for 7-10 days or until blood counts recover. Treatment repeats every 4 weeks for up to 12 courses.

NOTE: * Alternatively, patients may receive a single dose of pegfilgrastim SC, administered 48 hours after the completion of chemotherapy

Patients with intraocular lymphoma also receive methotrexate intravitreally twice weekly until the vitreous is clear of cells by slit lamp exam; once weekly for 1 month; and then monthly for 1 year.

Quality of life is assessed at baseline, every 3 months during treatment, within 30 days of final treatment, then every 6 months for 1 year, and then annually thereafter.

Patients are followed monthly for 3 months, every 2 months for 8 months, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 11-25 patients will be accrued for this study within 7-10 years.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed informed consent form in accordance with institutional guidelines
* Histologically or cytologically confirmed primary CNS lymphoma documented by brain biopsy or cerebrospinal fluid or vitrectomy analysis
* CD20 positive disease
* Progressive or relapsed disease during or after completion of prior methotrexate-based chemotherapy
* Aged 18 months to 75 years
* Performance status ECOG 0-3 OR Karnofsky 30-100%
* Hematocrit at least 25% (transfusion or epoetin alfa allowed)
* Absolute granulocyte count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3 OR at least lower limit of normal
* Bilirubin no greater than 2.0 times upper limit of normal
* Creatinine less than 1.8 mg/dL
* Calculated Creatinine clearance (CrCl) at least 50 mL/min
* Adequate cardiac function to tolerate general anesthesia
* Adequate pulmonary function to tolerate general anesthesia
* Available for follow-up for 1 year post therapy
* Fertile patients must use effective contraception for a minimum of 2 months before and during study participation

EXCLUSION CRITERIA:

* Radiographic signs of intra-cranial herniation and/or spinal block
* HIV positive
* Systemic lymphoma
* Positive serum HCG, pregnant or lactating
* Allergy to study agents
* Hepatitis B or hepatitis C positive

Ages: 18 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Good Samaritan Hospital Cancer Treatment Center, Hatton Institute, Cincinnati, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab and Carboplatin: Rituximab: (i.v.) 375 mg/m^2 given the evening before blood brain barrier disruption(BBBD) procedure day 1 Carboplatin: (i.a.) 200 mg/m^2 /day x 2 days = 400 mg/m^2
Period: Overall Study
Arm/Group | Rituximab and Carboplatin
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.235 (12.799)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response Rate to Chemotherapy Regimen Assessed by Radiographic Response at 2 Years.
Description: Per RECIST criteria (v1.1) and assessed by magnetic resonance imaging (MRI): Complete response (CR), Disappearance of all target lesions.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 17
Participants | 1

2. Secondary Outcome: Number of Participants With Overall Survival Assessed by Clinical and Radiographic Response
Description: Overall survival is measured from entry onto study until death from any cause or until death or progression of disease, respectively.
Time Frame: 5 years
Population: Data not collected due to low accrual and early termination.
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival Assessed by Clinical and Radiographic Response From First Day of Treatment Until Tumor Progression
Time Frame: 5 years
Population: Data not collected due to low accrual and early termination.
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life Assessed by EORTC QOL Before Treatment and Then Every 3 Months
Time Frame: 5 years
Population: Data not collected due to low accrual and early termination.
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Ototoxicity Assessed by Audiology Hearing Test Done Monthly During Treatment
Time Frame: 2 years
Population: Data not collected due to low accrual and early termination.
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 0

6. Secondary Outcome: Effect of Sodium Thiosulfate (STS) on Granulocytes and Erythrocytes Assessed by Complete Blood Count Lab Values Done Weekly During Treatment
Time Frame: 2 years
Population: Data not collected due to low accrual and early termination.
Arm/Group | Rituximab and Carboplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During study treatment (1 year).
Description: Unanticipated Problems (UP) and Adverse Events (AE) were reported to IRB according to OHSU's (coordinating center) policies, procedures and guidelines posted on the OHSU IRB web site. NCI Common Toxicity Criteria used to assess AEs.
Arm/Group | Rituximab and Carboplatin
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 16/17
Other Adverse Events (participants affected / at risk) | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab and Carboplatin (N=17)
Neutropenic Fever (Blood and lymphatic system disorders) | 2
Unresponsiveness (General disorders) | 1 — Hospitalized for unresponsiveness
Anemia (Blood and lymphatic system disorders) | 1
Superficial Epidermolysis (Musculoskeletal and connective tissue disorders) | 1
Neurological Symptoms (Psychiatric disorders) | 1
Stroke (Vascular disorders) | 1
Chemical Meningitis and Seizures (Vascular disorders) | 1
Extended Hospitalization (Investigations) | 2
Hospitalized for Fall (Injury, poisoning and procedural complications) | 1
Death (General disorders) | 1
Carotid Artery Tear (Blood and lymphatic system disorders) | 1
Electrolyte Imbalance and Increased Blood Sodium (Blood and lymphatic system disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab and Carboplatin (N=17)
Leg Pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No